CLINICAL TRIAL: NCT05153499
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial of the Efficacy, Safety, and Tolerability of a Single Oral Administration of CP101 for the Prevention of Recurrent Clostridioides Difficile Infection (CDI)
Brief Title: A Trial of CP101 for the Prevention of Recurrent CDI (PRISM4)
Acronym: PRISM4
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The termination of FIN-CDI-301 (PRISM4) is based on the voluntary, business-related decision of the sponsor.
Sponsor: Finch Research and Development LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FIN-CDI-301
Record Dates: First submitted 2021-11-17; First posted 2021-12-10 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Recurrent C. Difficile Infection
Keywords: C. difficile infection; recurrent Clostridium difficile infection; Clostriodioides difficile infection; recurrent C. diff infection; multiple recurrent C. diff infection; CDI; c. diff; microbiota transplantation; FMT; Fecal microbiota transplantation; Fecal microbiota transplant; Fecal transplant
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CP101 (Active Comparator)
  Interventions: Biological: CP101
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CP101 — CP101 is an investigational microbiome therapeutic designed to deliver a complete and functional microbiome to durably repair intestinal dysbiosis, which is being evaluated for the prevention of recurrent Clostridioides difficile infection (CDI).
  Arms: CP101
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial of the Efficacy, Safety, and Tolerability of a Single Oral Administration of CP101 for the Prevention of Recurrent Clostridioides difficile Infection (PRISM4). This Phase 3 trial will be conducted in 2 parts: a randomized, double-blind, placebo-controlled trial arm and an optional open-label treatment arm. After completing standard-of-care (SOC) CDI antibiotics for their most recent CDI recurrence, patients who meet all eligibility requirements will be randomized in a 2:1 ratio to receive either CP101 or placebo. Patients will be evaluated for CDI recurrence and safety follow-up through Week 8, the primary endpoint, as well as through Week 24. Patients who qualify may enroll into the optional open label arm if they experience CDI recurrence through week 8.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Men or women over 18 years of age or older
* Current diagnosis of a recurrence of non-severe, non-complicated CDI
* Subject has a clinical response to standard-of-care CDI antibiotics for the most recent CDI episode
* History of recurrent CDI defined as:

  * ≥ 3 episodes of CDI, with 2 episodes occurring within the previous 6 months (inclusive of the current episode); OR
  * Patients with a history of 2 episodes of CDI occurring within the previous 6 months (inclusive of the current episode) may be eligible if 65 years of age or older.
* For the Qualifying CDI episode, the following criteria must be satisfied:

  * History of diarrhea (> 3 unformed stools per day) for 2 or more consecutive days that is clinically consistent with CDI. AND
  * Documented positive stool test by local laboratory for toxigenic C. difficile (toxin enzyme immunoassay [EIA] or polymerase chain reaction [PCR]-based testing) for the current CDI episode and within 45 days prior to Randomization. AND
  * Received a course of SOC CDI antibiotics for the most recent CDI episode (for 10 to 21 days, with exact duration, antibiotic type, and dose at the discretion of the Investigator). AND
  * Demonstrated an adequate clinical response, defined as ≤ 3 unformed stools in 24 hours for 2 or more consecutive days during SOC CDI antibiotics prior to Randomization.

Exclusion Criteria:

* Known stool sample testing positive for enteric pathogen(s) (e.g., Salmonella, Shigella, diarrhoeagenic E. coli, Campylobacter, Giardia) within 28 days prior to Screening
* Pregnant, breast-feeding, or planning to become pregnant during the trial
* Historical or current diagnosis of inflammatory bowel disease
* Recent diagnosis (<6 months prior to screening) of diarrhea-predominant irritable bowel syndrome (post-infection or non-related to an enteric infection)
* Initiation of any systemic cancer treatment (e.g., chemotherapy, radiotherapy, biologic, immunotherapy, others) for active malignancy
* Major intra-abdominal surgery (e.g., bowel resection)
* Known primary or secondary immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (68):
- United States (61):
  - Mayo Clinic, Phoenix, Arizona
  - Facey Medical Foundation, Mission Hills, California
  - Kaiser Permanente Division of Research, Oakland, California
  - UCSF, San Francisco, California
  - Stanford Healthcare, Stanford, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Medical Research Center of Connecticut LLC, Hamden, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Christiana Care Health System, Newark, Delaware
  - George Washington University School of Medicine and Health, Washington D.C., District of Columbia
  - University of Florida Health, Gainesville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - ENCORE Borland-Groover Clinical Research, Jacksonville, Florida
  - San Marcus Research Clinic Inc, Miami, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Reliant Medical Research, Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Theia Clinical Research, LLC, St. Petersburg, Florida
  - Guardian Angel Research, Tampa, Florida
  - St Joseph's Comprehensive Research Institute, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - Metro Infectious Disease Consultants, Burr Ridge, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Iowa Clinic, Des Moines, Iowa
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Brigham and Womens Hospital, Boston, Massachusetts
  - William Beaumont Hospital, Farmington Hills, Michigan
  - Henry Ford Health System, Novi, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - MedPharmics LLC, Gulfport, Mississippi
  - St. Charles Clinical Research, LLC, Weldon Spring, Missouri
  - Mercury Street Medical Group, Butte, Montana
  - North Shore University Hospital-(Manhasset), Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Digiovanna Institute For Medical Education and Research, North Massapequa, New York
  - Central New York Research Corporation, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Brody School of Medicine at ECU, Greenville, North Carolina
  - Pinehurst Medical Clinic Inc, Pinehurst, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Gastro Health LLC, Cincinnati, Ohio
  - TruCare Internal Medicine & Infectious Diseases, DuBois, Pennsylvania
  - Regional GI, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Guthrie Clinic, Sayre, Pennsylvania
  - Women's Medicine Collaborative, Providence, Rhode Island
  - Lowcountry Infectious Diseases PA, Charleston, South Carolina
  - Main Street Physicians Care, Loris, South Carolina
  - Digestive Health Associates of Texas, PA, Carrollton, Texas
  - Kelsey Seybold Clinic, Houston, Texas
  - 1960 Family Practice P.A., Houston, Texas
  - Southern Star Research Institute LLC, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Infectious Diseases Associates of Central Virginia, Lynchburg, Virginia
- Canada (7):
  - University of Calgary - Calgary Health Region, Calgary, Alberta
  - CARe Clinic, Red Deer, Alberta
  - Yazdan Medical Corporation, Vancouver, British Columbia
  - Vancouver Island Health Authority, Victoria, British Columbia
  - Dalhousie University, Halifax, Nova Scotia
  - Saint Joseph's Health Care London, London, Ontario
  - University Health Network, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- CP101: CP101: CP101 is an oral investigational microbiome therapeutic designed to deliver a complete and functional microbiome to durably repair intestinal dysbiosis, which is being evaluated for the prevention of recurrent CDI.
- Placebo: Placebo: Matching placebo capsule
Period: Overall Study
Arm/Group | CP101 | Placebo
Started | 12 | 7
Completed | 4 | 2
Not Completed | 8 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Clinical Hold | 1 | 0
Not completed — Study Termination | 6 | 5

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population used.
Groups:
- Total: Total of all reporting groups
Arm/Group | CP101 | Placebo | Total
Number analyzed (Participants) | 12 | 7 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (14.8) | 66.6 (15.3) | 65.2 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 7 | 0 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 10 | 7 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 7 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Sustained Clinical Cure Through Week 8
Description: No data displayed because Outcome Measure has zero participants analyzed.
Time Frame: Week 8
Population: Study was terminated prematurely; data on primary endpoint are not available; therefore no analysis was conducted because there was no data to analyze.
Arm/Group | CP101 | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Sustained Clinical Cure Through Week 24
Description: No data displayed because Outcome Measure has zero participants analyzed.
Time Frame: Week 24
Population: Study was terminated prematurely; no data on secondary endpoint were available; therefore the analysis was not conducted because there are no data to analyze.
Arm/Group | CP101 | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: CDI Recurrence Through Week 24 as Evidenced by Positive Toxin EIA or Positive Toxigenic Culture
Description: No data displayed because Outcome Measure has zero participants analyzed.
Time Frame: Week 24
Population: Study was terminated prematurely; EIA testing was not performed on samples collected; therefore the analysis was not conducted because no data was available to analyze.
Arm/Group | CP101 | Placebo
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Improvement of Intestinal Microbiome Diversity at Week 1 as Determined by 16S Ribosomal Ribonucleic Acid (rRNA) Gene Amplicon Sequencing
Description: No data displayed because Outcome Measure has zero participants analyzed.
Time Frame: Week 1
Population: Study was terminated prematurely; Microbiome sample testing was not performed; therefore the analysis was not conducted because no data were available to analyze.
Arm/Group | CP101 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for a minimum of 30 days following treatment. Due to the early termination of the study, the longest follow-up period was 232 days.
Arm/Group | CP101 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/7
Other Adverse Events (participants affected / at risk) | 8/12 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CP101 (N=12) | Placebo (N=7)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural Haemotoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CP101 (N=12) | Placebo (N=7)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early. Most analyses were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restrictions on the PI are: (i) the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of up to twenty-four months from the lock-down of all study data and (ii) the sponsor can require the removal of its confidential information from results communications and may delay release for a period of up to 60 days for the purpose of filing patent applications.

DOCUMENTS (1):
  • Study Protocol (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT05153499/Prot_000.pdf